CLINICAL TRIAL: NCT04477096
Title: Study on the Drug Interaction of HS-10234 and Emtricitabine in Healthy Subjects
Brief Title: Evaluation of Drug Interaction Between HS-10234 and Emtriccitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HS-10234-108
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
Keywords: HIV
MeSH Terms: interventions — Emtricitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm for each part: two arms (Other): PART1:In the first period, HS-10234 will be administered at 25 mg QD for 7 days. In the second period, HS-10234 at 25 mg in combination with Emtricitabine at 200 mg will be administered QD for 7 days.
  PART2:In the first period, Emtricitabine will be administered at 200 mg QD for 7 days. In the second period, HS-10234 at 25 mg in combination with Emtricitabine at 200 mg will be administered QD for 7 days.
  Interventions: Drug: HS-10234; Drug: Emtricitabine

INTERVENTIONS:
Drug: HS-10234 — HS-10234
Drug: Emtricitabine — Emtricitabine

SUMMARY:
The study is being conducted to evaluate drug interaction between HS-10234 and Emtricitabine after multiple dose in healthy subjects.

DETAILED DESCRIPTION:
The study includes two parts. Part 1 is to evaluate the impact of Emtricitabine on HS-10234. Part 2 is to evaluate the impact of HS-10234 on Emtricitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent before any activities related to this trial and understand the procedures and methods of this trial;
2. Aged between 18 and 55 years old (including cutoff value), both male and female;
3. Male body weight ≥50.0kg, female body weight ≥45.0kg, body mass index (BMI) is 19~26 kg/m2 (including both ends);
4. Those who signed the informed consent form and had no birth plan within 3 months after the last dose and agreed to take effective contraceptive measures.

Exclusion Criteria:

1. People who have been or are currently suffering from any clinically serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities, or any other diseases that can interfere with the test results, Or have a stomach problem or have a history of stomach problems;
2. People who have drugs (penicillin or cephalosporin drugs), food, or have a history of allergy to test drugs or similar drugs;
3. If the subject have a history of surgery within the 4 weeks prior to the trial or plan to undergo surgery during the study period or have surgery that affected the absorption, distribution, metabolism, and excretion of drugs;
4. Those who took any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 14 days before taking the study drug, or those who were within 5 half-lives of the drug at the time of screening; those who plan to take non-study drugs or health products during the trial;
5. Those who participated in any drug clinical trial and used any trial drug within 3 months before administration (subject to the informed consent);
6. Participate in blood donation within 3 months before administration and the amount of blood donation >200 mL, or have received blood transfusion;
7. Unable or unwilling to follow the lifestyle guidelines required in the plan;
8. Smokers or those who smoked more than 5 cigarettes per day in the 3 months before the trial;
9. Alcoholics or frequent drinkers within 6 months before the test, that is, drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) or before administration Alcohol screening positive;
10. People who have a history of drug abuse, drug dependence, or a positive drug screen before administration;
11. Screening/baseline visit to alanine aminotransferase and/or aspartate aminotransferase and/or alkaline phosphatase and/or total bilirubin exceeds 1.2 times the upper limit of normal;
12. Abnormal vital signs (systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure <50 mmHg or >90 mmHg; pulse <50 bpm or >100 bpm) or physical examination, electrocardiogram, laboratory examination, imaging examination, etc. Abnormality has clinical significance (subject to the judgment of the clinical research doctor);
13. The QT interval is prolonged during screening (calculated using Bazett's method, male>450 msec, female>460 msec);
14. Hepatitis B surface antigen, hepatitis C antibody, syphilis serotonin, HIV antibody test positive;
15. Women during pregnancy or lactation;
16. Subjects may not be able to complete the study for other reasons or the investigator believes that they should not be included.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of HS-10234 and it's metabolite tenofovir, Emtricitabine | 0 - 24 hour on 7th day
  Cmax
Pharmacokinetics parameters of HS-10234 and it's metabolite tenofovir, Emtricitabine | 0 - 24 hour on 7th day
  AUC0-tau

SECONDARY OUTCOMES:
Concentration of HS-10234's metabolite tenofovir-diphosphate in peripheral blood mononuclear cells. | 0 - 24 hour on 7th day
  Concentration
Incidence of AEs, | 0 - 23 day
  laboratory abnormalities (based on hematology, biochemistry, and urinalysis tests)
Incidence of AEs, | 0 - 23 day
  body temperature
Incidence of AEs, | 0 - 23 day
  respiratory rate
Incidence of AEs, | 0 - 23 day
  blood pressure
Incidence of AEs, | 0 - 23 day
  pulse rate
Incidence of AEs, | 0 - 23 day
  Resting 12-lead ECG parameters（ECG QT Interval）

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Luo Y, Chen W, Yang G, Zou C, Huang J, Kuang Y, Shen K, Zhang B, Yang S, Xiang H, Li Z, Pei Q. Study on Pharmacokinetic Interactions Between HS-10234 and Emtricitabine in Healthy Subjects: An Open-Label, Two-Sequence, Self-Controlled Phase I Trial. Infect Dis Ther. 2022 Feb;11(1):175-186. doi: 10.1007/s40121-021-00555-y. Epub 2021 Oct 30. PMID 34727366